CLINICAL TRIAL: NCT04523831
Title: A Phase III Trial to Promote Recovery From Covid 19 With Combined Doxycycline and Ivermectin Along Standard Care
Brief Title: Clinical Trial of Ivermectin Plus Doxycycline for the Treatment of Confirmed Covid-19 Infection
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Dhaka Medical College (Other)
Responsible Party: Principal Investigator, Dr. Reaz Mahmud, Assistant Professor, Dhaka Medical College
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ERC-DMC/ECC/2020/117
Record Dates: First submitted 2020-08-19; First posted 2020-08-24 (Actual); Results first posted 2020-10-09 (Actual); Last update posted 2020-10-09 (Actual); Status verified 2020-10

CONDITIONS: Covid19
Keywords: Covid-19, Ivermectin
MeSH Terms: conditions — COVID-19 | interventions — Ivermectin; Doxycycline; imidazoleacetic acid; Standard of Care

STUDY DESIGN:
Intervention Model Description: Patient will be randomized 1:1 to placaebo with standard care and combined doxycycline and ivermectin with standard care.
Who Masked: Participant, Investigator
Masking Description: Double blind (The participant and the clinicians/data collectors will be unaware of the treatment the participant receives).The drugs will be labelled with a random code number
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ivermectin and Doxycycline (Active Comparator): Ivermactin 6 mg 2 tab stat, cap Doxycycline 100 mg 1 cap BD 5 days
  Interventions: Drug: Ivermectin and Doxycycline; Drug: Standard of care
- Placebo (Placebo Comparator): Standard treatment
  Interventions: Drug: Standard of care

INTERVENTIONS:
Drug: Ivermectin and Doxycycline — Ivermectin 6 mg, 2 tab stat and Doxycycline 100 mg twice daily for 5 days
  Other Names: Imac and Doxibac
  Arms: Ivermectin and Doxycycline
Drug: Standard of care — Paracetamol, Vitamin D, Oxygen if indicated, Low molecular weight heparin, dexamethasone if indicated

SUMMARY:
On 31 December 2019, the World Health Organization (WHO) was formally notified about a cluster of cases of pneumonia in Wuhan City, China. On 7 January the responsible virus was isolated and its genome sequence was shared on 12 January. It was named as COVID-19, a novel Coronavirus, SARS-CoV-2. It is a member of the Corona virus family which is RNA enveloped viruses.

Very rapidly the virus emerged as pandemic. Now it is dominating the lives of every people of this universe. Management of the COVID-19 relies on mainly supportive care and oxygen supplementation via non-invasive or mechanical ventilation in critical cases. Patients who are critically ill may also require vasopressor support and antibiotics for secondary bacterial infections.

There is no vaccine or highly effective antiviral drugs for COVID-19. Currently there is a tremendous effort around the world to develop effective preventive and therapeutic treatment for this disease.

World Health Organization has launched a non-blinded clinical trial (SOLIDARITY) to evaluate four candidate treatments (remdesivir, lopinavir/ritonavir, lopinavir/ritonavir/ interferon beta-1a, and chloroquine or hydroxychloroquine) versus standard of care in 18 countries worldwide. RECOVERY trial one of the largest trials to see the efficacy and safety of hydroxychloroquine revealed that they are no clear cut clinical benefit for COVID-19. Other drugs in the SOLIDARTY trial are quite expansive for resource limited countries like Bangladesh.

Study Published in the American Journal of Tropical Medicine advocates further research into Ivermectin for COVID-19 Treatment. The spotlight on Ivermectin was brought by Australian researchers from Monash University who demonstrated its efficacy against the SARS-CoV-2 coronavirus in vitro studies.

In different study Doxycycline also showed promising results in treatment of COVID 19 infection. It is highly lipophilic antibiotics that are known to chelate zinc component of matrix metalloprotienases (MMP). Corona viruses are known to rely heavily of MMPs for survival, cell infiltration and replication. It also has an anti-inflammatory effect which might be effective in combating cytokine storm of Covid-19 infection.

So it have been planned to conduct an experimental clinical trial using combination of ivermectin and doxycycline for treatment of COVID 19 along with the other standard care.

DETAILED DESCRIPTION:
OBJECTIVES:

General objectives:

To observe the benefit (clinical and microbiological) of Ivermectin and Doxycycline in Confirmed Covid 19 cases.

Specific objectives:

1. To observe the clinical outcome in trial group and the placebo group.
2. To observe the duration require controlling viral replication (negative RT-PCR) in the trial and placebo group.
3. To compare the outcome between the two groups.

RATIONALE:

Covid-19 is an emergent pandemic, threatens the life of millions of the people throughout the globe. There is increasing effort of the scientist to unveil a remedy of covid-19. Still it is unsuccessful. At present there is no other alternative other than experimenting the existent drug against the virus. There are several trials going throughout the globe. Among them Ivermectin showed good efficacy in vitro trial. Some clinical trial also proved it beneficial. The Doxycycline also has some anti viral role with its prominent anti-inflammatory role. Synergistic action of the two drugs might be proved some benefit in clinical trial. As both drugs are cheap and less toxic, if it does, it would be the blessing for the poor people of the globe.

METHODOLOGY:

Study type: Interventional Clinical trial Estimated enrollment: 200 participants per group

For superior trial, the formula is:

N=size per group; p=the response rate of standard treatment group; p0= the response rate of new drug treatment group; zx= the standard normal deviate for a one or two sided x; d= the real difference between two treatment effect; δ0= a clinically acceptable margin; S2= Polled standard deviation of both comparison groups.

All parameters were assumed as follows: p =0.40; p0=0.58; α=0.05;β=0.20; δ=0.18; δ0=0.10.

However, we are assuming that lost to follow up or refuse to include in trial will be 20%, that means 24. So at least 150 patients will be allocated randomly and power of this study will be 80%.

Allocation: Randomized Intervention model: Parallel assignment Intervention model description: Patient will be randomized 1:1 to placaebo with standard care and combined doxycycline and ivermectin with standard care.

Blinding: Double blind (The participant and the clinicians/data collectors will be unaware of the treatment the participant receives) Primary purpose: Treatment Official title: A phase III trial to promote recovery from covid 19 with combined Doxycycline and Ivermectin along standard care. Provider of placebo and active ingredients: Popular pharmaceutical limited Dosage of the drugs: Ivermactin 6 mg 2 tab stat, cap Doxycycline 100 mg 1 cap BD 5 days

Data collection technique:

Data will be collected by assigned. trained data collectors (Physician). Patient will be enrolled according to defined inclusion and exclusion criteria in the current research. Informed written consent will be obtained from the patient or their relatives. Each patient participating in the trial will be uniquely identified, and information such as his name, address is recorded in the trial 'subject number list'. Only the principle investigator will be aware about the allocation of the drugs. The patients and the data collectors will be unaware about the group allocation of the drugs. The Data will be reviewed by the co-investigators. It will be managed by principle and co-principle investigators in designated computer.

Clinical assessment (fever, cough, Anorexia, Temperature, pulse, blood pressure, respiratory rate, oxygen saturation) will be done every day. Routine investigation (CBC, ESR, CRP, Creatinine, RBS, SGPT, chest x-ray, D- Dimer) will be done at admission and at day 3, 5, 7, 10 and 14 day. In case of the clinical deterioration it would done according to necessity. RT-PCR will be done at day-0, Day 5, day 7 and day 14.

Standard care: both the experimental and placebo will receive the available standard of care, like-

* Paracetamol, Antihistamine, Cough suppressant, Vitamins
* Oxygen therapy according to indication and need
* Low molecular weight heparin according to indication
* Appropriate other broad spectrum antibiotics
* Other drugs for associated co- morbid condition

Management of the adverse events:

Drugs adverse effect will be monitored by a defined committee. The patient experiencing adverse effect of the drugs will be discontinued from the study. It will be managed with priority to the highest possible level by the hospital authority as well as the investigators.

If the patient progresses from mild to moderate or severe disease, the study will be continued and available management of the appropriate severity will be immediately started. The patient will be monitored closely.

Data analysis:

Data will be analyzed by computer with the help of SPSS (Statistical Package for Social Sciences) version 26. Unpaired t-test would be used for testing quantitative data and for testing qualitative data two sample z- test will be used. Comparing drug outcome in between two groups hazard ratio, Kaplan-Meire curve will be used.

Dropout management: Likelihood based methods such as mixed models will be used to estimate unbiased treatment effects, under assumptions regarding the missingness mechanisms.

ELIGIBILITY:
Inclusion Criteria:

* COVID-19 infection, confirmed by polymerase chain reaction (PCR) test within 3 days from enrollment
* Only mild and moderate COVID-19 infected cases
* Able to provide informed consent

Exclusion Criteria:

* Unable to take oral medication
* Pregnant or breast feeding lady
* Patients with severe COVID symptoms or admission in ICU/HDU
* Alanine Aminotransferase (ALT) or aspartate aminotransferase (AST) more than 5 upper limit of normal (ULN)
* On non-invasive positive pressure ventilation or mechanical ventilation at time of study entry
* Known hypersensitivity to Doxycycline or ivermectin or its components.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2020-08-22 (Actual); Study Completion 2020-09-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mahmud Reaz, FCPS, Principal Investigator — Assistant Professor
Locations (1):
- Dhaka Medical College, Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: Yes
Patients age, sex, Date of covid positive report, Symtoms,Date of covid negative report, post covid symptoms, time to recover.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: September 2020 to December 2020
Access Criteria: Person who are investigating covid-19 in various aspects

REFERENCES:
- [Derived] Mahmud R, Rahman MM, Alam I, Ahmed KGU, Kabir AKMH, Sayeed SKJB, Rassel MA, Monayem FB, Islam MS, Islam MM, Barshan AD, Hoque MM, Mallik MU, Yusuf MA, Hossain MZ. Ivermectin in combination with doxycycline for treating COVID-19 symptoms: a randomized trial. J Int Med Res. 2021 May;49(5):3000605211013550. doi: 10.1177/03000605211013550. PMID 33983065

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was designed to evaluate the effects of potential treatments in hospitalized and outdoor patients with mild to moderate COVID-19 infection, from 1 June to 30 august, 2020 in the largest COVID-19 dedicated hospital, Dhaka Medical College Hospital in Bangladesh.
Pre-assignment Details: Of 556 patients who screened and were assessed for eligibility, 400 underwent randomization. Total 200 patients received active drug and 200 patient received placebo.
Groups:
- Ivermectin and Doxycycline: Ivermactin 6 mg 2 tab stat, cap Doxycycline 100 mg 1 cap BD 5 days
  Ivermectin and Doxycycline: Ivermectin 6 mg stat and Doxycycline 100 mg twice daily for 5 days
Period: Overall Study
Arm/Group | Ivermectin and Doxycycline | Placebo
Started | 200 | 200
Completed | 183 | 180
Not Completed | 17 | 20
Not completed — Lost to Follow-up | 15 | 17
Not completed — Death | 0 | 3
Not completed — Adverse Event | 2 | 0

BASELINE CHARACTERISTICS:
Population: We followed intention to treat analysis; SPSS (Statistical Package for Social Sciences) version 20 was used to analyze data. To compare mean of the two group chi square test was done.
Groups:
- Total: Total of all reporting groups
Arm/Group | Ivermectin and Doxycycline | Placebo | Total
Number analyzed (Participants) | 200 | 200 | 400
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.72 (14.28) | 38.47 (11.89) | 39.59 (13.17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 77 | 88 | 165
  Male | 123 | 112 | 235
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Early Clinical Improvement
Description: Number of patients have clinical improvement as described by WHO and Bangladesh local guideline with 7 days..
  1. Body temperature remains normal for at least 3 days (ear temperature is lower than 37.5 °C).
  2. Respiratory symptoms are significantly improved.
  3. Lung imaging shows obvious improvement in lesions.
  4. There is no co-morbidities or complications which require hospitalization.
  5. SpO2, >93% without assisted oxygen inhalation.
Time Frame: 7 days
Population: Intention to treat analysis. Linear logistic regression
Measure: Count of Participants; unit: Participants
Groups:
- Ivermectin Plus Doxycycline: Ivermectin plus Doxycycline plus Standard of care
- Placebo: Placebo plus Standard of care
Arm/Group | Ivermectin Plus Doxycycline | Placebo
Number analyzed (Participants) | 183 | 180
Participants | 111 | 80
Statistical Analysis 1: Comparison: Ivermectin Plus Doxycycline vs Placebo; Test type: Superiority; p < 0.03, Regression, Linear; Cox Proportional Hazard = 0.53, 95% CI 2-sided [0.30 to 0.96]

2. Primary Outcome: Number of Participants With Late Clinical Recovery
Description: Number of the patients required more than 12 days for clinical improvement as defined above.
Time Frame: 12 days
Population: Intention to treat analysis. Binary logistic regression
Measure: Count of Participants; unit: Participants
Arm/Group | Ivermectin Plus Doxycycline | Placebo
Number analyzed (Participants) | 183 | 180
Participants | 42 | 67
Statistical Analysis 1: Comparison: Ivermectin Plus Doxycycline vs Placebo; Test type: Superiority; p < 0.004, Regression, Logistic; Cox Proportional Hazard = 0.51, 95% CI 2-sided [0.32 to 0.80]

3. Secondary Outcome: Number of Patients Having Clinical Deterioration.
Description: Number of patients deteriorating to next level of severity, like moderate, severe and death. That is from mild illness at presentation with subsequent follow up developed moderate, severe illness or death. Like wise from moderate illness at presentation developed severe illness or death.
  Mild illness: These patients usually present with symptoms of an upper respiratory tract viral infection, including mild fever, cough (dry), sore throat, nasal congestion, malaise, headache, muscle pain, or malaise. Signs and symptoms of a more serious disease, such as dyspnea, are not present Moderate illness: Respiratory symptoms such as cough and shortness of breath (or tachypnea in children) are present without signs of severe pneumonia.
  Severe illness:severe dyspnea, respiratory distress, tachypnea (> 30 breaths/min), and hypoxia (SpO2 < 90% on room air).
Time Frame: 1 month
Population: Intention to treat analysis. Binary Logistic regression
Measure: Count of Participants; unit: Participants
Groups:
- Ivermectin Plus Doxycycline: Ivermection plus Doxycycline Plus standard of Care
Arm/Group | Ivermectin Plus Doxycycline | Placebo
Number analyzed (Participants) | 183 | 180
Participants | 16 | 32
Statistical Analysis 1: Comparison: Ivermectin Plus Doxycycline vs Placebo; Test type: Superiority; p < 0.013, Regression, Logistic; Cox Proportional Hazard = 0.45, 95% CI 2-sided [0.23 to 0.85]

4. Secondary Outcome: Number of Patients Remain Persistently Positive for RT-PCR of Covid-19
Description: Number of Patients remain positive for RT-PCR of Covid-19 at day 14 after the day of initial positivity.
Time Frame: 14 days
Population: Intention to treat analysis. Binary logistic regression
Measure: Count of Participants; unit: Participants
Arm/Group | Ivermectin Plus Doxycycline | Placebo
Number analyzed (Participants) | 183 | 180
Participants | 14 | 36
Statistical Analysis 1: Comparison: Ivermectin Plus Doxycycline vs Placebo; Test type: Superiority; p < 0.001, Regression, Logistic; Cox Proportional Hazard = 0.58, 95% CI 2-sided [0.44 to 0.81]

ADVERSE EVENTS:
Time Frame: 1 month
Groups:
- Ivermectin and Doxycycline: Ivermectin Plus Doxycycline plus standard of care
Arm/Group | Ivermectin and Doxycycline | Placebo
All-Cause Mortality (participants affected / at risk) | 0/183 | 3/180
Serious Adverse Events (participants affected / at risk) | 2/183 | 0/180
Other Adverse Events (participants affected / at risk) | 7/183 | 0/180
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ivermectin and Doxycycline (N=183) | Placebo (N=180)
Erosive esophagitis (Gastrointestinal disorders) | 2 (2) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 3.8% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ivermectin and Doxycycline (N=183) | Placebo (N=180)
Non ulcer Dyspepsia (Gastrointestinal disorders) | 7 (7) | 0 (0)

LIMITATIONS AND CAVEATS:
We followed up the patients by telephonic (video) interview, which has some inherent drawback for the study. we could not assess viral clearance directly. Only single dose regimen was used. Efficacy might higher if the different regimen would use.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol and Informed Consent Form (2020-08-26): https://cdn.clinicaltrials.gov/large-docs/31/NCT04523831/Prot_ICF_000.pdf
  • Statistical Analysis Plan (2020-08-26): https://cdn.clinicaltrials.gov/large-docs/31/NCT04523831/SAP_001.pdf